CLINICAL TRIAL: NCT07184905
Title: Effect of Oral Bifidobacterium Longum on Skin Barrier Dysfunction in Obesity: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Oral Bifidobacterium Longum for Skin Barrier Dysfunction in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LL-KY-2025110-02
Record Dates: First submitted 2025-08-06; First posted 2025-09-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Skin Barrier to Water Loss; Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral administration of inactive Bifidobacterium longum group (Sham Comparator)
  Interventions: Biological: Oral administration of inactive Bifidobacterium longum group
- Oral Bifidobacterium longum group (Experimental)
  Interventions: Biological: Oral Bifidobacterium longum group

INTERVENTIONS:
Biological: Oral administration of inactive Bifidobacterium longum group — 1×10^11 CFU of inactive Bifidobacterium longum was given orally once daily for one month
  Arms: Oral administration of inactive Bifidobacterium longum group
Biological: Oral Bifidobacterium longum group — 1×10^11 CFU of Bifidobacterium longum was given orally once daily for one month
  Arms: Oral Bifidobacterium longum group

SUMMARY:
This clinical trial aims to evaluate the safety and efficacy of oral Bifidobacterium longum supplementation for treating obesity-induced skin barrier impairment in individuals aged 18-40 with BMI ≥30, compared to healthy controls. The study focuses on the following questions:

Can oral Bifidobacterium supplementation reduce skin barrier damage (measured by transepidermal water loss/TEWL) in obese participants? Does modulation of gut microbiota with Bifidobacterium longum impact skin barrier function and systemic inflammation?

Researchers will compare outcomes across two groups:

* Intervention Group (Obese): Oral Bifidobacterium longum capsules
* Placebo Control Group (Obese): Oral inactive Bifidobacterium longum (heat-killed)

Participant Procedures:

Take daily oral capsules (Bifidobacterium longum or inactive strain) for 4 weeks Undergo non-invasive skin testing (TEWL measurements) at baseline and study completion Provide blood, stool, and skin swab samples for inflammation and microbiome analyses Complete weekly check-ins to report adverse effects (e.g., gastrointestinal discomfort, skin irritation)

ELIGIBILITY:
Inclusion Criteria :

* 1. Meets 2020 WHO BMI classification:
* a. Normal weight (18.5-24.9 kg/m²)
* b. Overweight (25-29.9 kg/m²)
* c. Obesity (≥30 kg/m²)
* 2. Presence of skin barrier impairment (e.g., dryness, erythema, desquamation, or itching)
* 3. Age 18-40 years
* 4. Generally good health (no active systemic diseases)
* 5. Able and willing to provide written informed consent
* 6. No use of oral/topical medications or probiotics within 6 months prior
* 7. No active skin disease or traumatic skin lesions

Exclusion Criteria :

* 1. Known allergy or hypersensitivity to probiotics, placebo, or investigational product
* 2. Active skin disease (e.g., psoriasis, eczema, infection) requiring treatment
* 3. Severe medical conditions:
* a. Cardiopulmonary disease (NYHA class III/IV)
* b. Uncontrolled diabetes (HbA1c >9%)
* c. Autoimmune disorders
* 4. Pregnant or breastfeeding women
* 5. Any condition that may interfere with protocol compliance (per investigator judgement), including:
* a. Inability to understand study procedures
* b. History of poor clinical trial adherence
* 6. Concurrent participation in other interventional trials

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Mean change in transepidermal water loss (TEWL, g/h/m²) on the volar forearm from baseline to 1 month after intervention, measured by Tewameter | Baseline through 1 month after intervention
  TEWL will be assessed on the volar aspect of the forearm using a Tewameter device under standardized environmental conditions (controlled temperature and humidity). At each time point, TEWL will be measured at three predefined skin sites on the volar forearm, and the average value will be used. The primary outcome will be the mean change in TEWL (g/h/m²) from baseline (Day 0) to 1 month after intervention. Lower TEWL values indicate improved skin barrier function.

SECONDARY OUTCOMES:
Change in gut Bifidobacterium longum abundance and metabolites in fecal samples | Baseline through 1 month after intervention
  Stool samples will be collected at baseline and after intervention. Microbial abundance will be assessed by 16S rRNA sequencing, and metabolites will be profiled using targeted metabolomics. Data will be reported as relative abundance (%) and metabolite concentrations (µM).
Change in serum inflammatory cytokine levels | Baseline through 1 month after intervention
  Serum samples will be collected before and after Bifidobacterium longum treatment. Cytokine levels (e.g., IL-6, TNF-α, IL-22) will be measured by ELISA, reported as pg/mL.
Change in skin hydration measured by Corneometer | Baseline through 1 month after intervention
  Skin hydration will be assessed using a Corneometer device. Outcomes will be expressed as mean skin capacitance values (arbitrary units) at baseline and post-intervention.
Change in clinical skin health score | Baseline through 1 month after intervention
  Skin dryness, scaling, erythema, itching, and allergy-related symptoms will be evaluated using a standardized Skin Dryness Scoring System. Data will be reported as mean score change from baseline.
Change in body weight and BMI | Baseline through 1 month after intervention
  Participants' body weight (kg) and BMI (kg/m²) will be recorded at baseline and post-intervention. Data will be reported as mean change.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No